CLINICAL TRIAL: NCT00109031
Title: A Randomized, Blinded, Active-control Trial of Palifermin (rHuKGF) to Evaluate Oral Mucositis in Subjects With Hematologic Malignancies Undergoing Fractionated Total Body Irradiation (fTBI) and High Dose Chemotherapy With Autologous Peripheral Blood Progenitor Cell (PBPC) Transplantation
Brief Title: Palifermin for the Reduction of Oral Mucositis in Single-dose Evaluation (PROMISE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20040212; NCT00126529 (obsolete NCT alias); NCT00965692 (obsolete NCT alias)
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Cancer; Lymphoma; Leukemia
Keywords: Cancer; Oncology
MeSH Terms: conditions — Neoplasms; Lymphoma; Leukemia | interventions — Fibroblast Growth Factor 7; Whole-Body Irradiation; Cyclophosphamide; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Palifermin 60 µg/kg for 3 days (Active Comparator): Palifermin 60 µg/kg plus placebo to match the total volume equivalent to a 180 µg/kg dose on the 3 days prior to fractionated total body irradiation (fTBI) and palifermin 60 µg/kg on Days 0, 1 and 2 after peripheral blood progenitor cell transplantation (PBPC). Participants also received conditioning therapy with fTBI and cyclophosphamide/etoposide prior to PBPC transplantation on Day 0.
  Interventions: Drug: palifermin; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Placebo
- Palifermin 180 μg/kg on Day -1 (Experimental): Palifermin 180 μg/kg on Day -1 and matched placebo on Days -2 and -3 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC. Participants also received conditioning therapy with fTBI and cyclophosphamide/etoposide prior to PBPC transplantation on Day 0.
  Interventions: Drug: palifermin; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Placebo
- Palifermin 180 μg/kg on Day -2 (Experimental): Palifermin 180 μg/kg on Day -2 and placebo on Days -1 and -3 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC. Participants also received conditioning therapy with fTBI and cyclophosphamide/etoposide prior to PBPC transplantation on Day 0.
  Interventions: Drug: palifermin; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Placebo
- Palifermin 180 μg/kg on Day -3 (Experimental): Palifermin 180 μg/kg on Day -3 and placebo on Days -1 and -2 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC. Participants also received conditioning therapy with fTBI and cyclophosphamide/etoposide prior to PBPC transplantation on Day 0.
  Interventions: Drug: palifermin; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Placebo

INTERVENTIONS:
Drug: palifermin — Administered as one daily intravenous bolus.
  Other Names: Kepivance; Recombinant Human Keratinocyte Growth Factor (rHuKGF)
Radiation: Total Body Irradiation — To be delivered before the administration of chemotherapy in 6, 8, or 10 fractions over 3 or 4 days.
Drug: Cyclophosphamide — Cyclophosphamide is administered at a total dose of 100 mg/kg given in 1 dose on Day -2
Drug: Etoposide — Etoposide may be administered (optional) as a single intravenous infusion over 4 hours on the day after the last fTBI fraction.
  Other Names: VP-16
Drug: Placebo — Administered as one daily intravenous bolus.

SUMMARY:
To evaluate whether palifermin (rHuKGF) administered as a single dose is non-inferior to 3 consecutive doses of palifermin in reducing the incidence of severe oral mucositis (World Health Organization [WHO] grade 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Subjects with: non-Hodgkin's lymphoma, Hodgkin's disease, acute myelogenous leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, chronic lymphocytic leukemia, or multiple myeloma
* Minimum of 1.5 x 10^6 CD34+ cells/kg cryopreserved and to be transplanted.

Exclusion Criteria:

* Cancer other than those specified in inclusion criteria above (except: adequately treated basal cell carcinoma of the skin)
* Prior bone marrow or peripheral blood stem cell transplantation - Negatively selected (purged) stem cell product - Current active infection or oral mucositis
* Congestive heart failure as defined by New York Heart Association class III or IV.
* History of or current diagnosis of pancreatitis
* Inadequate renal function (serum creatinine greater than 1.5x the upper limit of normal per the institutional guidelines)
* Inadequate liver function (direct bilirubin greater than 1.5x the upper limit of normal, aspartate aminotransferase (AST) greater than 3x upper limit of normal and/or alanine aminotransferase (ALT) greater than 3x upper limit of normal per the institutional guidelines)
* Inadequate pulmonary function as measured by a corrected diffusion capacity of carbon monoxide (DLCO) less than 50% of predicted.
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-01; Primary Completion 2006-02 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Started | 11 | 10 | 14 | 12
Completed | 11 | 8 | 12 | 12
Not Completed | 0 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Primary Analysis Set (all randomized participants who signed informed consent before invasive, protocol-specified procedures).
Groups:
- Palifermin 60 µg/kg for 3 Days: Palifermin 60 µg/kg on the 3 days prior to fractionated total body irradiation (fTBI) and palifermin 60 µg/kg on Days 0, 1 and 2 after peripheral blood progenitor cell transplantation (PBPC).
- Palifermin 180 μg/kg on Day -1: Palifermin 180 μg/kg on Day -1 and placebo on Days -2 and -3 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC.
- Palifermin 180 μg/kg on Day -2: Palifermin 180 μg/kg on Day -2 and placebo on Days -1 and -3 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC.
- Palifermin 180 μg/kg on Day -3: Palifermin 180 μg/kg on Day -3 and placebo on Days -1 and -2 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC.
- Total: Total of all reporting groups
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3 | Total
Number analyzed (Participants) | 11 | 10 | 13 | 12 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.9) | 49.7 (9.7) | 47.4 (14.2) | 46.1 (13.8) | 48.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 4 | 2 | 11
  Male | 6 | 10 | 9 | 10 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 11 | 8 | 12 | 10 | 41
  Black or African American | 0 | 2 | 1 | 1 | 4
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
Type of diagnosis [Number; unit: participants] — Acute lymphoblastic leukemia., Acute myelogenous leukemia, Chronic lymphocytic leukemia, and1 ( 8) Chronic myelogenous leukemia are subsets of Leukemia.
  participants
    Hodgkin's disease | 0 | 1 | 4 | 4 | 9
    Non-Hodgkin's lymphoma | 9 | 9 | 9 | 6 | 33
    Multiple Myeloma | 0 | 0 | 0 | 0 | 0
    Leukemia | 2 | 0 | 0 | 2 | 4
    Acute lymphoblastic leukemia | 1 | 0 | 0 | 0 | 1
    Acute myelogenous leukemia | 1 | 0 | 0 | 1 | 2
    Chronic lymphocytic leukemia | 0 | 0 | 0 | 1 | 1
    Chronic myelogenous leukemia | 0 | 0 | 0 | 0 | 0
Etoposide use [Number; unit: participants]
  Yes | 9 | 10 | 11 | 11 | 41
  No | 2 | 0 | 2 | 1 | 5
Number of days of total body irradiation [Number; unit: participants] — Data are reported for the safety analysis set, as treated. Seven participants received the wrong sequence of placebo and palifermin in error in. Consequently, 10, 11, 13, and 12 participants actually received treatment according in each treatment arm respectively.
  participants
    ≤ 2 days | 0 | 1 | 1 | 0 | 2
    3 days | 4 | 4 | 6 | 4 | 18
    4 days | 6 | 6 | 6 | 8 | 26
    ≥ 5 days | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Oral Mucositis (WHO Grade 3 and 4)
Description: Participants underwent evaluations of oral mucosal (OM) surfaces (mucositis assessments) daily during hospitalization and daily thereafter until severe OM returned to grade ≤ 2. A trained evaluator documented the findings using the World Health Organization (WHO) oral toxicity scale according to the following: Grade 0 = None; Grade 1 = Soreness, erythema; Grade 2 = Erythema, ulcers, ability to eat solids; Grade 3 = Ulcers, requires liquid diet; Grade 4 = Alimentation not possible.
Time Frame: Up to Day 28
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Number analyzed (Participants) | 11 | 10 | 13 | 12
participants
  Yes | 9 | 6 | 4 | 9
  No | 2 | 3 | 9 | 3
  Missing | 0 | 1 | 0 | 0

2. Secondary Outcome: Duration of Severe Oral Mucositis (WHO Grade 3 and 4)
Description: The duration of severe oral mucositis (OM) was calculated as the number of days from the onset of severe OM (first time a WHO grade 3 or 4 was observed) to the day when severe OM was resolved (first time WHO grade 2 or less was observed after last WHO grade 3 or 4). Durations of 0 days were assigned to those participants who did not experience any WHO grade 3 or 4 during the study.
Time Frame: Up to Day 28
Population: Primary analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Number analyzed (Participants) | 11 | 10 | 13 | 12
days | 6.0 (4.1) | 4.4 (5.4) | 1.9 (3.6) | 5.1 (4.1)

3. Secondary Outcome: Area Under the Curve (AUC) of Mouth and Throat Soreness Score
Description: The Oral Mucositis Daily Questionnaire (OMDQ) is a self-reported tool that evaluates overall health, mouth and throat soreness (MTS) and activity limitations due to MTS. The OMDQ was completed once daily beginning with the first day of study drug administration through Day 28. The area under the curve of mouth and throat soreness score was assessed from the question "How much mouth and throat soreness did you experience in the past 24 hours?" Participants answered on a scale from 0 (no soreness) to 4 (extreme soreness). A higher value in MTS AUC indicates worse self-assessed MTS.
Time Frame: From the first day of study drug administration through Day 28
Population: Primary analysis set with available MTS data
Measure: Mean (Standard Deviation); unit: MTS score * days
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Number analyzed (Participants) | 11 | 10 | 13 | 11
MTS score * days | 26.4 (22.4) | 45.1 (14.4) | 30.4 (18.6) | 30.9 (16.1)

4. Secondary Outcome: Number of Participants With Parenteral or Transdermal Opioid Analgesic Use
Description: Includes nonprophylactic intravenous opioid analgesics (fentanyl, morphine, morphine sulphate, hydromorphone, meperidine) and transdermal opioid analgesics (fentanyl patch) for the indication of oral mucositis and dysphagia.
Time Frame: Up to Day 28
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Number analyzed (Participants) | 11 | 10 | 13 | 12
participants
  Yes | 7 | 7 | 7 | 9
  No | 4 | 3 | 6 | 3

5. Secondary Outcome: Number of Participants With WHO Grades 2, 3 or 4 Oral Mucositis
Description: Participants underwent evaluations of oral mucosal (OM) surfaces (mucositis assessments) daily during hospitalization and daily thereafter until OM returned to grade ≤ 2. A trained evaluator documented the findings using the World Health Organization (WHO) oral toxicity scale according to the following: Grade 0 = None; Grade 1 = Soreness, erythema; Grade 2 = Erythema, ulcers, ability to eat solids; Grade 3 = Ulcers, requires liquid diet; Grade 4 = Alimentation not possible.
Time Frame: Up to Day 28
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Number analyzed (Participants) | 11 | 10 | 13 | 12
participants
  Yes | 10 | 8 | 9 | 12
  No | 1 | 1 | 4 | 0
  Missing | 0 | 1 | 0 | 0

6. Secondary Outcome: Duration of WHO Grade 2, 3 or 4 Oral Mucositis
Description: The duration of grade 2, 3 or 4 oral mucositis (OM) was calculated as the number of days from the onset of grade 2, 3 or 4 OM (first time a WHO grade 2, 3 or 4 was observed) to the day when WHO grade 2 - 4 OM was resolved (first time WHO grade less than 2 was observed after last WHO grade 2, 3 or 4). Durations of 0 days were assigned to those participants who did not experience any WHO grade 2, 3 or 4 during the study.
  OM was evaluated using the World Health Organization (WHO) oral toxicity scale according to the following: Grade 0 = None; Grade 1 = Soreness, erythema; Grade 2 = Erythema, ulcers, ability to eat solids; Grade 3 = Ulcers, requires liquid diet; Grade 4 = Alimentation not possible.
Time Frame: Up to Day 28
Population: Primary analysis set with available OM assessment data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Number analyzed (Participants) | 11 | 9 | 13 | 12
days | 10.3 (4.9) | 9.0 (8.2) | 4.7 (4.2) | 9.4 (5.7)

7. Secondary Outcome: Number of Participants With WHO Grade 4 Oral Mucositis
Description: as for outcome 5
Time Frame: Up to Day 28
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Palifermin 60 µg/kg for 3 Days | Palifermin 180 μg/kg on Day -1 | Palifermin 180 μg/kg on Day -2 | Palifermin 180 μg/kg on Day -3
Number analyzed (Participants) | 11 | 10 | 13 | 12
participants
  Yes | 5 | 5 | 2 | 3
  No | 6 | 4 | 11 | 9
  Missing | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 40 days from first dose of palifermin
Description: Seven participants received the wrong sequence of placebo and palifermin as follows (# participants [from assigned arm to actual treatment arm]): 2 participants (A to C), 2 participants (D to B), 1 participant (C to A), 1 participant (B to D), 1 participant (C to D). Adverse event data are summarized by actual treatment group.
Groups:
- Palifermin 60 µg/kg for 3 Days (A): Palifermin 60 µg/kg on the 3 days prior to fractionated total body irradiation (fTBI) and palifermin 60 µg/kg on Days 0, 1 and 2 after peripheral blood progenitor cell transplantation (PBPC).
- Palifermin 180 μg/kg on Day -1 (B): Palifermin 180 μg/kg on Day -1 and placebo on Days -2 and -3 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC.
- Palifermin 180 μg/kg on Day -2 (C): Palifermin 180 μg/kg on Day -2 and placebo on Days -1 and -3 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC.
- Palifermin 180 μg/kg on Day -3 (D): Palifermin 180 μg/kg on Day -3 and placebo on Days -1 and -2 prior to fTBI, and palifermin 60 μg/kg on Days 0, 1, and 2 after PBPC.
Arm/Group | Palifermin 60 µg/kg for 3 Days (A) | Palifermin 180 μg/kg on Day -1 (B) | Palifermin 180 μg/kg on Day -2 (C) | Palifermin 180 μg/kg on Day -3 (D)
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/11 | 4/13 | 1/12
Other Adverse Events (participants affected / at risk) | 9/10 | 10/11 | 12/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin 60 µg/kg for 3 Days (A) (N=10) | Palifermin 180 μg/kg on Day -1 (B) (N=11) | Palifermin 180 μg/kg on Day -2 (C) (N=13) | Palifermin 180 μg/kg on Day -3 (D) (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Engraftment syndrome (Immune system disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin 60 µg/kg for 3 Days (A) (N=10) | Palifermin 180 μg/kg on Day -1 (B) (N=11) | Palifermin 180 μg/kg on Day -2 (C) (N=13) | Palifermin 180 μg/kg on Day -3 (D) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 3 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 8 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 5 | 8 | 6
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral mucosal discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Tongue geographic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 5 | 5 | 6
Asthenia (General disorders) | 2 | 2 | 3 | 2
Axillary pain (General disorders) | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 1 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 2 | 1 | 2 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 6 | 2 | 5 | 5
Feeling jittery (General disorders) | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 2 | 0 | 4
Oedema peripheral (General disorders) | 1 | 3 | 3 | 1
Pain (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 3 | 2 | 1
Tenderness (General disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Engraftment syndrome (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 2
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 2
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Delayed engraftment (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gingival injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 1 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 5 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 3 | 4 | 1
Headache (Nervous system disorders) | 2 | 3 | 3 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Unresponsive to verbal stimuli (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 6 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 2 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 2 | 2
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 5
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 6 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 3 | 3 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.